CLINICAL TRIAL: NCT04147104
Title: ecco2R to facilitatE earLy libEration From mechanicAl Ventilation inpatientS With Copd Acute Exacerbation
Acronym: RELEASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Quiron Sagrado Corazon (Other)
Responsible Party: Principal Investigator, Luis Morales, MD, Hospital Quiron Sagrado Corazon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/53-UCI-HUSC
Record Dates: First submitted 2019-10-27; First posted 2019-10-31 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Acute Exacerbation of COPD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care plus invasive mechanical ventilation (Active Comparator): Invasive mechanical ventilation for lung support and to facilitate exhalation via an endotracheal tube o tracheotomy.
  Interventions: Device: Invasive mechanical ventilation
- ECCO2R plus invasive mechanical ventilation (Experimental): Low-flow ECCO2R adjunct to standard-of-care and invasive mechanical ventilation.
  Interventions: Device: Low flow ECCO2R; Device: Invasive mechanical ventilation

INTERVENTIONS:
Device: Low flow ECCO2R — Treatment with a medical device called ECCO2R. The device consists of a drainage cannula placed in a large central vein, a membrane lung (artificial gas exchanger), and a return cannula into the venous system. Blood is pumped through the membrane lung, and CO2 is removed by diffusion. A flowing gas known as "sweep gas" containing little or no CO2 runs along the other side of the membrane, ensuring a diffusion gradient from blood to the other side, hence promoting CO2 removal.
  Arms: ECCO2R plus invasive mechanical ventilation
Device: Invasive mechanical ventilation — Invasive mechanical ventilation deviceto support acute respiratory failure and facilitate exhalation via an endotracheal tube or tracheotomy.

SUMMARY:
A pragmatic randomised controlled trial to determine whether early Veno-Venous Extracorporeal Carbon Dioxide Removal (VV-ECCO2R) in mechanically ventilated patients with acute exacerbated Chronic Obstructive Pulmonary Disease decreases the days of invasive mechanical ventilation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major worldwide health burden. Currently, it is the fourth leading cause of death worldwide, and is the only leading cause of death that is rising, and will likely become the third cause of death by 2020. COPD is characterized by progressive destruction in the elastic tissue within the lung, causing respiratory failure.

Patients with COPD may experience acute exacerbations with severe hypercapnic respiratory failure. Hypercapnia results from acute worsening of expiratory flow limitation caused by the increased small airway resistance with consequent development of dynamic alveolar hyperinflation and intrinsic positive end-expiratory pressure (PEEP). In the most severe cases, these may be refractory to conventional therapies and mechanical ventilation, becoming life-threatening.

Extracorporeal carbon dioxide removal (ECCO2R) represents an attractive approach in this setting. The last decade has seen an increasing interest in the provision of extracorporeal support for respiratory failure, as demonstrated by the progressively increasing number of scientific publications on this topic. In particular, remarkable interest has been focused on extracorporeal carbon dioxide removal (ECCO2R), due to the relative ease and efficiency in blood CO2 clearance granted by extracorporeal gas exchangers as compared to oxygen delivery.

In recent years, a new generation of ECCO2R devices has been developed. More efficient veno-venous (VV)-ECCO2R devices have become available and have replaced the arterio-venous approach, having the advantage of not requiring arterial puncture.

The new VV-ECCO2R devices offer lower resistance to blood flow, have smaller priming volumes, and provide a much more efficient gas exchange with relatively low extracorporeal blood flows (0.4-1 L/min). The technology of these devices is now comparable to that of renal dialysis and has been experimented in several animal and human studies, demonstrating a significant reduction in arterial CO2 and improvement in the work of breathing.

In summary, minimally invasive ECCO2R appears very promising for patients with acute exacerbation of obstructive diseases refractory to conventional treatment, but systematic evaluation is needed to prove its clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Age ≥ 18
  * Known or suspected aeCOPD that failed NIV that requires invasive mechanical ventilation
  * Failed treatment with NIV defined as:
* NIV for at least 2 hours and no more than 24 hours with signs of respiratory distress (respiratory rate > 30 breaths/min and use of accessory muscles or paradoxical abdominal movements) AND
* PaCO2> 55 mmHg and pH < 7.25 or pH < 7.30 and PaCO2 > 55 mmHg, with PaCO2 decrease < 20% from baseline

  • Known or suspected aeCOPD patients where NIV is contraindicated and need immediate invasive mechanical ventilation due to:
* Respiratory arrest
* Inability to protect the airway (impaired cough or swallowing or massive aspiration or respiratory pauses with loss of consciousness or gasping of air)
* Inability to clear secretions
* Agitated and confused patients
* Facial deformities or conditions that prevent mask from fitting
* Uncooperative or unmotivated patients

Exclusion Criteria:

* Participation in other interventional studies
* Patients already included in this study that need a new readmission because of a new aeCOPD episode
* aeCOPD intubated > 12 hours
* Extubation within the previous 48 hours following intubation and invasive mechanical ventilation due to any cause
* Anatomical abnormalities or vascular diseases preventing the correct insertion of the ECCO2R cannula
* PaO2 to FiO2 ratio < 150 on PEEP ≥ 5 cmH2O
* Known or suspected pregnancy (women of childbearing potential require a pregnancy test)
* Hemodynamic instability defined as

  * MAP < 60 mmHg despite the infusion of fluids or vasoactive drugs OR
  * Failure to increase systolic blood pressure above 80-90 mmHg OR
  * Need for inotropic drugs to maintain systolic blood pressure> 85 mmHg OR
  * ECG evidence of ischemia or significant uncontrolled ventricular arrhythmia
* Acute multiple organ failure defined as more than two organ failures assessed by SOFA score. Organ dysfunction can be identified as an acute change in total SOFA score > 2 points
* Decompensated heart failure defined as an exacerbation of symptoms or signs after a period of relative stability such as dyspnea, fatigue or edema in the setting of previously established myocardial dysfunction (systolic or diastolic)32 and B-natriuretic peptide more than100 ng/L.
* Tracheostomized patients
* Untreated pulmonary embolism, pleural effusion, pneumothorax or bronchopleural fistula as the primary cause of acute respiratory failure
* Hemoglobin < 7 gr/dL that require daily transfusion to maintain hemoglobin above 7 gr/dL at the time of screening
* Active major bleeding defined as35:

  * Fatal bleeding
  * Bleeding that is symptomatic and occurs in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, pericardial, in a non-operated joint, or intramuscular with compartment syndrome, assessed in consultation with the MD
  * Extrasurgical site bleeding causing a fall in hemoglobin level of 2 gr/dL or more or leading to transfusion of two or more units of whole blood or red cells, with temporal association within 24-48 hours to the bleeding
* Recent major surgery in the last 2 weeks
* Platelet count < 50 000/mm3
* Prothrombin time-international normalized ratio (INR) > 1.5 in the absence of anticoagulation therapy
* Heparin-induced thrombocytopenia (HIT) or known paradoxical/allergic reactions to heparin
* History within the previous 3 months of stroke or severe head trauma or intracranial arterio-venous malformation, or cerebral aneurysm, or central nervous mass lesion or intracranial bleeding
* Epidural catheter in place or plan to insert an epidural catheter during the study
* Gastrointestinal bleeding within the 6 weeks prior to study entry
* Severe liver insufficiency (Child-Pugh scores >7) or INR > 1.6 suspected to be related to liver disease (liver associated coagulopathy)
* Presence of severe (acute or chronic) renal failure defined as requiring any form of dialysis (including CRRT and CVVH) and/or having a serum creatinine > 2.5 mg/dL and urine clearance < 20 mL/hour
* Inability to receive blood products
* History of complications from extracorporeal support
* Permanent home ventilation except for sleep-disordered breathing
* Significant weakness or paralysis of respiratory muscles due to causes unrelated to aeCOPD
* Recent (< 7 days) prolonged (> 24 hours) use of muscle paralyzing agents
* Immunocompromised state defined as

  * Received chemotherapy or radiation within the previous 45 days and still under treatment for the underlying cancer
  * Received or currently receiving immunosuppressive therapy, excluding corticosteroids, within the last 3 months
  * Known to have AIDS defined illness
* Patients not expected to survive 6 months on the basis of premorbid health status
* History of uncontrolled, major psychiatric disorder
* Therapeutic restriction (DNR), moribund patient or not expected to survive current hospitalization
* Consent declined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The amount of time in the first 28 days following randomization that a patient is free of ventilatory support including non-invasive ventilation | 28 days
  Statistically analyzed as Ventilator-Free Days during the 28 days from randomization (VFD-28)

SECONDARY OUTCOMES:
All-cause (health-related) mortality at 28 and 90 days from randomization | 28 and 90 days
  Incidence of health-related deaths at 28 and 90 days from randomization, regardless of subject location at time of death.
Health-related quality of life (HRQoL) | 90 days after randomization
  EQ-5D-5L is a generic preference-based measure of health, which provides a description of health using five dimensions (mobility, self-care, usual activities, pain/discomfort and anxie-ty/depression) each with 5 levels of severity.
Catheter-related complications | Participants will be followed for the duration of ICU stay, an expected average of 30 days
  Bleeding, malposition, dislodgement or kinking, infection, vascular occlusion, thrombosis, hematoma, aneurism, pseudoaneurysm formation
Work of breathing | Participants will be followed for the duration of ICU stay, an expected average of 4 days
  Assessed by respiratory rate (cutoff 30 breaths/min) and use of accessory muscles or paradoxical abdominal movements
Time to ECCO2R cessation | Participants will be followed for the duration of ICU stay, an expected average of 4 days
  Defined as from the onset of ECCO2R to 6 hours following cessation of CO2 removal
Length of ECCO2R in situ | 7 days
  Defined as the insertion of cannulas until there removal
Time to normalization of pH and PaCO2 | 3 hours
Length of ICU stay | 4 days
  Participants will be followed for the duration of ICU stay
Hospital Length of stay | 10 days
  Participants will be followed for the duration of hospital stay
Incidence of new tracheostomies | Within 28 days from randomization
  Incidence of new tracheostomies
Tolerance of ECCO2R therapy | 4 days
  Assessed by comfort, defined according a visual analog comfort scale (VAS). The VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best).
Dyspnea | 4 days
  Assessed by the modified Borg scale. This is a scale rates the difficulty of breathing. It starts at number 0 where dyspnea is causing no difficulty at all and progresses through to number 10 where dyspnea is maximal.
ICU Mobility | Randomization to end of treatment or 14 days, whichever is sooner
  Ability of subject to mobilize in bed and out of bed while in Intensive Care as assessed using ICU Mobility Score (IMS)
Incidence of failed extubations | Within 28 days from randomization
  Incidence of re-intubation within 48 hours of extubation for original exacerbation
Frailty Index Score | 90 days after randomization
  The Clinical Frailty Scale is scored on a scale from 1 (very fit) to 9 (terminally ill) and is based on clinical judgment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Artigas, MD, Principal Investigator — Hospital Universitari Sagrat Cor, Grupo Quironsalud

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access request will be reviewed by an External Independent Review Panel. Requestors will be required to signed a Data Access.

REFERENCES:
- [Background] Del Sorbo L, Pisani L, Filippini C, Fanelli V, Fasano L, Terragni P, Dell'Amore A, Urbino R, Mascia L, Evangelista A, Antro C, D'Amato R, Sucre MJ, Simonetti U, Persico P, Nava S, Ranieri VM. Extracorporeal Co2 removal in hypercapnic patients at risk of noninvasive ventilation failure: a matched cohort study with historical control. Crit Care Med. 2015 Jan;43(1):120-7. doi: 10.1097/CCM.0000000000000607. PMID 25230375
- [Background] Burki NK, Mani RK, Herth FJF, Schmidt W, Teschler H, Bonin F, Becker H, Randerath WJ, Stieglitz S, Hagmeyer L, Priegnitz C, Pfeifer M, Blaas SH, Putensen C, Theuerkauf N, Quintel M, Moerer O. A novel extracorporeal CO(2) removal system: results of a pilot study of hypercapnic respiratory failure in patients with COPD. Chest. 2013 Mar;143(3):678-686. doi: 10.1378/chest.12-0228. PMID 23460154